CLINICAL TRIAL: NCT06327477
Title: First-in-Human Phase I and II Study to Determine Safety and Efficacy of Proton-Spatially Fractionated Radiotherapy (P-SFRT) in Retroperitoneal Soft Tissue Sarcoma
Brief Title: Proton-Spatially Fractionated Radiotherapy and Standard Radiation Therapy for the Treatment of Newly Diagnosed Retroperitoneal Soft Tissue Sarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NU 23S01; NCI-2024-01927 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00220015; NU 23S01 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Retroperitoneal Sarcoma
MeSH Terms: interventions — Biopsy; Specimen Handling; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (P-SFRT, IG-IMRT) (Experimental): Patients undergo P-SFRT over 1 fraction and then undergo IG-IMRT over 25-28 fractions for 35 to 42 days. Patients undergo surgical resection 21 to 35 days after radiation therapy. Patients undergo blood sample collection during screening and on study. Patients also undergo biopsy during screening and CT on study and on follow up.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Resection; Radiation: Spatially-fractionated Radiation Therapy

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Radiation: Intensity-Modulated Radiation Therapy — Undergo IG-IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
Radiation: Spatially-fractionated Radiation Therapy — Undergo P-SFRT
  Other Names: GRID Therapy; SFRT

SUMMARY:
This phase I/II trial studies the side effects and best dose of proton-spatially fractionated radiotherapy (P-SFRT) and to see how well it works with standard radiation therapy in treating patients with newly diagnosed retroperitoneal soft tissue sarcoma. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Standard spatially fractionated radiotherapy (SFRT) refers to how the radiation is delivered to the tumor. SFRT means that different parts of the tumor are receiving different doses of radiation (fractionation) through beams that allow areas of higher and lower (peaks and valleys) of doses of the radiation. This spatial fractionation allows an overall high-dose radiation to be given in the peaks and those areas of the tumor may release cells and substances that may help with killing tumor cells, reducing tumor symptoms and shrinking tumors. Proton therapy is a type of radiation therapy that can overcome some of the barriers of standard SFRT. Protons are tiny radioactive particles that can be controlled in a beam to travel up to the tumor and, compared to the particles used in standard radiotherapy, proton therapy can deliver higher doses to the tumor because smaller doses of radiation are delivered to tissues away from the tumor. This allows radiation therapy dose-escalated (continuously increasing the dose of radiation) treatment to tumors even though the tumor is near radiation sensitive organs like the colon. Giving P-SFRT with standard radiation therapy may work better in treating patients with newly diagnosed retroperitoneal soft tissue sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) for P-SFRT, which will be used as the recommended phase II dose (RP2D) for P-SFRT prior to standard fractionated radiation therapy and surgical intervention for retroperitoneal sarcoma (RPS). (Phase I) II. To determine the efficacy of P-SFRT prior to standard fractionated radiation therapy and surgical intervention for RPS. (Phase II)

SECONDARY OBJECTIVES:

I. To determine whether P-SFRT is safe when administered prior to standard fractionated radiation therapy and surgery for RPS. (Phase I) II. To determine progression-free survival (PFS) in patients with RPS who have been treated with P-SFRT prior to standard fractionated radiation therapy and surgical intervention. (Phase II) III. To determine overall survival (OS) in patients with RPS who have been treated with P-SFRT prior to standard fractionated radiation therapy and surgical intervention. (Phase II) IV. To determine objective response (OR) in patients with RPS who have been treated with P-SFRT prior to standard fractionated radiation therapy and surgical intervention. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of P-SFRT followed by a phase II study.

Patients undergo P-SFRT over 1 fraction and then undergo image-guided intensity modulated radiation therapy (IG-IMRT) over 25-28 fractions for 35 to 42 days. Patients undergo surgical resection 21 to 35 days after radiation therapy. Patients undergo blood sample collection during screening and on study. Patients also undergo biopsy during screening and computed tomography (CT) on study and on follow up.

After completion of study treatment, patients are followed up at 30 and 90 days after surgery, and then up to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed, histologically or cytologically confirmed, untreated retroperitoneal soft tissue sarcoma
* The soft-tissue sarcoma tumor must be at least 3 cm in diameter
* Patients must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1.
* Patients must be age ≥ 18 years on day of signing any informed consent documents
* Patients must exhibit a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale or >70% on the Karnofsky Scale
* Leukocytes (white blood cells [WBC]) ≥ 3,000/mcL
* Absolute neutrophil count (ANC) ≥ 1,500/mcL

  * Note: growth factor/transfusion is not permitted prior to these measurements being taken
* Hemoglobin (Hgb) ≥ 9 g/d
* Platelets (PLT) ≥ 100,000/mcL
* Total bilirubin < 1.5 x upper limit of normal (ULN) (or direct bilirubin < ULN)
* Aspartate Transferase (AST) ( serum glutamic-oxaloacetic transaminase [SGOT]) ≤ 2.5 x institutional ULN
* Alanine transaminase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) ≤ 2.5 x institutional ULN
* Creatinine ≤ 1.5 x upper limit of normal (ULN)
* Creatinine clearance ≥ 50mL/min
* International normalized ratio (INR) (or prothrombin time [PT] or partial thromboplastin time [PTT]; one will be used) < 1.5 x ULN (unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants [within 10 days of treatment initiation])
* Activated partial thromboplastin time (aPTT) < 1.5 X ULN (unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants [within 10 days of treatment initiation])
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients of child-bearing potential (POCBP) must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) from time of informed consent and for the duration of study participation. Patients who can impregnate their partners must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) from time of informed consent and for the duration of study participation. Should a patient become pregnant or suspect they are pregnant while they or their partner is participating in this study, they should inform their treating physician immediately.

  * Note: At the discretion of the investigator, acceptable methods of contraception may include total abstinence in cases where the lifestyle of the patient ensures compliance. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
  * Note: A POCBP is any person with an egg-producing reproductive tract (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* POCBP must have a negative urine pregnancy test within 72 hours prior to undergoing CT simulation for P-SFRT. If a urine pregnancy test is positive or cannot be confirmed negative, a serum pregnancy test will be required
* POCBP must be willing and able to use an adequate method of contraception
* Patients with sperm-producing reproductive capacity (PWSPRC) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from time of informed consent, for the duration of study participation, and for 120 days following completion of therapy. PWSPRC treated or enrolled on this protocol must also agree to refrain from donating sperm from time of informed consent for the duration of study participation and for 120 days following completion of therapy
* Patients must have the ability to understand and the willingness to sign a written informed consent document
* Patients must be medically fit to undergo surgery
* Patients must have plans to undergo neoadjuvant radiation therapy and surgery with curative intent

Exclusion Criteria:

* Patients who have had one of the following soft tissue sarcoma subtypes where neoadjuvant chemotherapy is established as standard-of-care:

  * Extra-skeletal Ewing sarcoma
  * Embryonal rhabdomyosarcoma
  * Alveolar rhabdomyosarcoma
  * Desmoplastic small round cell tumor
* Patients who have had any prior radiation therapy to the affected area
* Patients who have had chemotherapy, radiotherapy, or other antineoplastic agents ≤ 28 days (6 weeks for nitrosureas or mitomycin C) prior to planned treatment start date
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who have taken steroid therapy or any other immunosuppressive therapy within 7 days of first dose prior to trial treatment
* Patients with a known history of active tuberculosis (TB) (Bacillus tuberculosis)
* Patients with a known history of active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected) infection
* Patients with current or a history of any distant metastatic disease (including brain). Note: an isolated or oligo-metastatic regional occurrence may be allowed if all other criteria have been met and curative attempt is being pursued
* Patients with a known history of (non-infectious) pneumonitis that required steroids or had evidence of current pneumonitis
* Patients who have received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally killed virus vaccines, and as such, patients who have received these vaccines are not excluded; however, intranasal influenza vaccines are live attenuated vaccines and are not allowed
* Patients who have had an allogenic tissue/solid organ transplant
* Patients with a history of inflammatory bowel disorders (i.e., ulcerative colitis, Crohn's disease) or rheumatologic disorders (i.e., Sjogren's, scleroderma, rheumatoid arthritis) that serve as a contraindication to retroperitoneal radiation therapy
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Major surgery within 30 days of registration
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient¡¦s safety or study endpoints
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Patients who are pregnant (positive urine pregnancy test within 72 hours prior to enrollment) or nursing. If a urine pregnancy test is positive or cannot be confirmed negative, a serum pregnancy test will be required
* Patients who are expecting to become pregnant or impregnate their partner within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Patients who are currently participating in or have participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Other study specific or disease criteria for exclusion (e.g., certain disease sub-types that are not eligible, patients who are unable to swallow oral medication if the study involves oral agents, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (Phase I) | Up to the first 30 days of treatment
  Will be defined as the highest dose with a dose-limiting toxicity (DLTs) as determined in phase I using Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0). The DLT will be considered toxic and the prior dose will be considered the MTD (maximum tolerated dose). For the purposes of this protocol, the MTD will be the recommended phase II dose (RP2D).
Pathological complete response (Phase II) | Up to 3 years
  Efficacy will be determined based on pathologic complete response (pCR). A pathologist will score the efficacy and the percentage necrosis which will be based on tissue samples removed during surgery or biopsy after treatment with radiation or chemotherapy.

SECONDARY OUTCOMES:
Incidence of adverse events (Phase I) | Up to 3 years
  Will be summarized by providing a frequency of adverse events (CTCAE v 5.0) by severity, type, timing, and attribution for toxicities of any grade, with rates of ≥ grade 3 toxicities also analyzed separately. Adverse event rates will be summarized and accompanied by 95% exact binomial CIs.
Overall response rate (ORR) (Phase II) | Assessed up to 3 years
  Using imaging, patients who experience an objective response (confirmed complete response [CR] or confirmed partial response [PR] per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1)].
Progression-free survival (PFS) (Phase II) | Assessed up to 3 years
  Will be assessed by disease progression and is defined as progressive disease (PD) per RECIST v 1.1, other documented clinical or radiographical progression per physician judgment, or death due to disease.
Overall survival (OS) ( (Phase II) | Assessed up to 3 years
  Overall survival will be calculated as the time that elapses between baseline (day of surgery) and the date of death from any cause for all evaluable patients.

CONTACTS AND LOCATIONS:
Overall Officials: Seth M Pollack, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States